CLINICAL TRIAL: NCT06386367
Title: Monastery-based Health Education by Buddhist Monks to Promote Malaria Knowledge and Preventive Practices in Rural Myanmar: A Quasi-experimental Study
Brief Title: Health Education by Buddhist Monks to Promote Malaria Knowledge and Preventive Practices in Rural Myanmar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Myanmar Health Network Organization (Other)
Collaborators: Chulalongkorn University (Other); Ministry of Health and Sports, Myanmar (Other Government)
Responsible Party: Principal Investigator, Pyae Linn Aung, Principal Investigator, Myanmar Health Network Organization
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MHNO-001
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Buddhist Monks; Health Education; Malaria; Monastery-based; Myanmar; Preventive Practice
MeSH Terms: conditions — Health Education; Malaria

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monastery-based health education intervention (Experimental): The education sessions were conducted in Burmese by trained monks. They followed the normal teachings of the Buddhist doctrine and typically lasted 30-40 minutes. Our research utilized Burmese as the medium for delivering health messages, and all accompanying materials were meticulously prepared in Burmese. The study team observed at least one to two education sessions in each study village.
  Interventions: Behavioral: Monastery-based health education by Buddhist monks
- Control (No Intervention): Participants in the control group just received routine malaria control services such as diagnostic, treatment and bed net distribution.

INTERVENTIONS:
Behavioral: Monastery-based health education by Buddhist monks — During the three-month intervention from July to September 2022, a total of 18 health education sessions were conducted across the three intervention villages, with an average of 50 attendees per session, totaling 921 attendees across all sessions.
  Arms: Monastery-based health education intervention

SUMMARY:
Malaria is still a leading public health concern in Myanmar. However, people living in rural areas usually showed poor prevention practice despite residing in malaria hotspots. The majority in Myanmar are Buddhists who frequently visit the monastery and receive the speech delivered by the monks. In a malaria high burden township of the Sagaing Region from northern Myanmar, current study will first explore the difference in malaria preventive practices among people residing in different malaria-endemic villages through a mixed-methods approach. Next, this research will address the knowledge gaps by a monastery-based health education delivered by trained Buddhist monks using standardized health messages instruction for six consecutive months between August 2022 to January 2023. To test whether the intervention could balance those gaps among different groups, quantitative data of baseline, 3-month, and 6-month will be compared using descriptive statistics, chi-square test, T-test or repeated ANOVA, and the Difference-In-Differences (DID) analysis, as applicable.

ELIGIBILITY:
Inclusion Criteria:

For educational intervention; - voluntary participation

For questionnaire surveys;

* male or female household leaders or immediate family members
* aged >18 years who had resided in the study villages for more than one year

Exclusion Criteria:

For questionnaire surveys;

- Individuals who were unable to communicate effectively or were under the influence of narcotics, including alcohol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 501 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Malaria knowledge and preventive practices | Pre intervention (July 2022), 3-month post-intervention (Dec 2022) and 6-month post-intervention (Mar 2023)
  To assess pre-existing malaria knowledge and preventive practices among both intervention and control groups, pre-intervention surveys were conducted. Subsequently, three- and six-month post-intervention surveys were conducted to evaluate changes following the intervention. A validated questionnaire translated from English to Burmese was used. The questionnaire comprised three sections: demographic information of the respondents, knowledge of malaria and preventive practices. Each section had multiple small questions, and each correct answer was scored. The resultant scores were aggregated, wherein every participant had the potential to accrue a maximum of ten points pertaining to the attribution of malaria causation, symptoms of malaria, and adoption of personal preventative measures against malaria. The participants were eligible to secure eight points in the domain of malaria diagnosis and treatment, alongside twelve scores for the use of LLINs.

CONTACTS AND LOCATIONS:
Locations (1):
- Myanmar Health Network Organization, Yangon, Burma

IPD SHARING:
Plan to Share IPD: Undecided